CLINICAL TRIAL: NCT06534346
Title: A Randomized, Open, Single-dose, Two-cycle, Two-sequence, Cross-over Design Phase I Clinical Study to Evaluate the Effect of Food on the Pharmacokinetic Profile of a Single Oral DA-302168S Tablet in Healthy Subjects
Brief Title: The Food Effect on Pharmacokinetics of DA-302168S
Acronym: DA168
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chendu DIAO Pharmaceutical Group CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-CP-DA168-04
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Single-dose clinical trial with healthy volunteers sequentially using a single dose of DA-302168S tablet under fasting and thereafter under fed conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-302168S (fed+fasting) (Experimental)
  Interventions: Drug: 15 mg DA-302168S tablet
- DA-302168S (fasting+fed) (Experimental)
  Interventions: Drug: 15 mg DA-302168S tablet

INTERVENTIONS:
Drug: 15 mg DA-302168S tablet — Qualified subjects will be randomly assigned to one of two dosing sequences in a 1:1 ratio. Either DA-302168S tablet with food on Day 1 and DA-302168S tablet without food on Day 6 (treatment sequence fed/fasted), or DA-302168S tablet without food on Day 1 and DA-302168S tablet with food on Day 6 (treatment sequence fasted/fed).
  Each administration sequence consists of two cycles, with one administration per cycle and a 5-day washout period between each administration.
  Other Names: DA168

SUMMARY:
This study will be conducted to determine the effect of food on the pharmacokinetics characteristic of DA-302168S following administration of a DA-302168S tablet with and without a high-fat meal.

DETAILED DESCRIPTION:
This study plans to enroll 16 participants. Qualified subjects will be randomly assigned to one of two dosing sequences (The first group will receive DA-302168S tablets on an fasting condition, followed by administration after high-fat meals. The second group adopts the opposite administration methods) in a 1:1 ratio. Each administration sequence consists of two cycles, with one administration per cycle and a 5-day washout period between each administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years old (including 18 and 55 years old), male or female.
* Weight: male ≥50kg, female ≥45kg, body mass index (BMI) in the range of 19.0 ~ 28.0kg/m2 (including the end value).
* Subjects and their spouses or partners did not plan to become pregnant or plan to donate sperm or ovum during the study period until 3 months after the last dose, and agreed to use at least one acceptable and effective contraceptive method
* Subjects and their spouses or partners did not plan to become pregnant or plan to donate sperm or eggs during the study period until 3 months after the last dose, and agreed to use at least one acceptable and effective contraceptive method.
* No clinically significant abnormalities identified in the judgement of investigator at screening.
* Written informed consent prior to any study specific procedures.

Exclusion Criteria:

* subjects with a history of abnormal clinical presentation, diseases to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, endocrine system, renal, hepatic, gastrointestinal, respiratory, metabolic, and skeletal systems, and a history of malignant tumors, which are judged to be clinically significant by the Investigator.
* Use of any medication (including prescription, over-the-counter, herbal, etc.) or nutraceutical within 14 days prior to the first dose.
* May have any contraindications, allergies or hypersensitivity to DA-302168S Tablets (both test drug and placebo) or its excipients, GLP-1RA, DPP-4 analogues.
* Previous family history of medullary thyroid carcinoma or type 2 multiple endocrine adenoma syndrome.
* History or evidence of any of the following conditions:

  1. decompensated heart failure (New York Heart Association (NYHA) Cardiac Classification III and IV [Appendix 5: NYHA Heart Failure Classification]), cardiac arrhythmias (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, second or third degree atrioventricular block, QTcF intervals > 450 milliseconds for men or > 470 milliseconds for women [Appendix 8: Fridericia Method Corrected QT Interval Formula], PR intervals > 220 milliseconds, etc.) prior to the first administration of the study drug. (e.g., supraventricular tachycardia, atrial fibrillation, atrial flutter, grade II or III AV block, QTcF interval >450 ms in males or >470 ms in females [Appendix 8: Formula for Correcting QT Intervals by the Fridericia Method], PR interval >220 ms, etc.) and who, in the opinion of the investigator, are unsuitable for participation in this study;
  2. Serious trauma or acute infection that may affect glycemic control within 4 weeks prior to screening;
  3. Positive results for any of the Hepatitis B Surface Antigen, Hepatitis C Antibody, Syphilis Spirochete Antibody, or Human Immunodeficiency Virus (HIV) Antibody;
  4. Mental or neurological illness prior to screening, unwillingness to communicate, or a language barrier that prevents full understanding and cooperation;
  5. Other medical or psychiatric conditions that may increase the risk of participation in the study or that, in the judgment of the Investigator, may make the subject unsuitable for participation in the study, including a recent history (within the past two years) of major depression or other serious mental disorder, or any history of attempted suicide.
* Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg prior to the first dose and who, in the opinion of the investigator, are not suitable for participation in the study.
* Those who screen positive for substance abuse or have a history of substance abuse within the past five years or have used drugs in the 3 months prior to screening.
* Those who have participated in a clinical trial of another drug within 3 months prior to screening and have received any of the clinical trial drugs.
* Elective surgery was planned during the study period.
* Those who have donated or lost ≥200mL of blood, received a blood transfusion, or used blood products within 3 months prior to screening.
* Female subjects are pregnant or lactating.
* Those who consumed excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day, or who consumed tea, coffee and/or caffeinated beverages within 48 hours prior to the first dose of the drug, or who were unable to discontinue consumption during the trial period
* Previous chronic intake of xanthine- or grapefruit-rich beverages or foods, or consumption of any xanthine- or grapefruit-rich product within 48 hours prior to the first dose.
* Smokers or those who smoked an average of ≥5 cigarettes per day in the 3 months prior to screening, or those who were unable to stop using any tobacco-based products during the trial.
* Heavy drinkers or regular drinkers in the 3 months prior to screening, i.e., those who consume more than 14 standardized units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of 40% alcohol by volume spirits or 150 mL of wine) or those who have a positive breath test for alcohol at baseline or who are unable to discontinue the use of any alcohol-containing product during the test period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
  Peak Plasma Concentration of DA-20168S
Tmax | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
  Tmax will be determined from the observed plasma concentration data.
AUC0-t AUC0-t | Days 1 and 6: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 and 72 hours postdose.
  AUC, calculated using linear up/ log down trapezoidal method from time zero to time t, where t is the time of the last measurable concentration.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | 13 days
  Incidence,duration and severity of adverse events according to NCI-CTCAE v5.0.
Concentration of blood glucose | Pre-dose and postdose on day 1 and day 6.
  Fasting and postprandial blood glucose will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Doctor, Principal Investigator — Gulou Hospital Affiliated to Nanjing Medical University, Jiangsu, China.
Locations (1):
- Gulou Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No